CLINICAL TRIAL: NCT01404871
Title: Predicting Medication Response in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Obsessive Compulsive Foundation (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Dr. Peggy Richter, Director, Clinic for OCD & Related Disorders Head, Frederick W. Thompson Anxiety Disorders Centre Dept. of Psychiatry, Sunnybrook Health Sciences Centre Associate Professor of Psychiatry, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: OCF-Richter
Record Dates: First submitted 2009-02-06; First posted 2011-07-28 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; pharmacogenetics; cortical inhibition; genetics
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Clomipramine; Escitalopram; Dexetimide; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomization to ECIT or CMI (Active Comparator): Randomized trial of clomipramine or escitalopram
  Interventions: Drug: clomipramine; Drug: escitalopram
- Open label Duloxetine (Active Comparator): Open label trial of duloxetine
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: clomipramine — oral tablets, starting at 50mg/daily for 12 weeks including > 8 weeks at 250 mg/daily
  Other Names: Anafranil
  Arms: Randomization to ECIT or CMI
Drug: escitalopram — oral tablet, starting 10mg/daily 12 week treatment including >8 weeks at max dose 50mg daily
  Other Names: Cipralex
  Arms: Randomization to ECIT or CMI
Drug: duloxetine — oral tablets, starting dose 30mg daily 12 week treatment including >8weeks at 120mg daily
  Other Names: Cymbalta
  Arms: Open label Duloxetine

SUMMARY:
In this study, the investigators hope to study a number of variables the investigators believe may help us predict why some people respond better to some medications than others. Participants will be randomly assigned to receive one of two typical medications for OCD, clomipramine or escitalopram. Individuals who would like to participate but who have previously tried one or both of these medications may instead take a newer drug, duloxetine, and undergo the identical procedures. The factors the investigators will be studying include demographics (i.e. age, gender, age of onset of OCD), genetic markers (such as variants in genes involved in breaking down drugs in the liver (cytochrome P450 system), and genes involved in several brain chemical systems, such as serotonin), the dimensions of OCD symptoms (i.e. checking, washing, and hoarding) and cortical inhibition. Cortical inhibition will be measured transcranial magnetic stimulation and is being studied because deficits in this process may be important in the development of OCD. The investigators hypothesize that certain pretreatment clinical characteristics will correlate with poor treatment response including earlier age of onset, longer duration of illness, increased YBOCS severity and presence of significant hoarding symptoms. The investigators expect that increasing degree of deficit in CI pre-treatment will predict poor treatment response, but that increase in CI from pre- to post-treatment will correlate with a positive treatment response. Differences in genetic marker status for cytochrome P450 genes will correlate with tolerability and/or response, as well as differences in genetic marker status in SLC1A1, GRIN2B, 5HT1B and 5HT2A will correlate with response.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Obsessive Compulsive Disorder
* Must be able to swallow tablets

Exclusion Criteria:

* History of stroke
* History of Parkinson's disease
* History of Epilepsy
* Clinical diagnosis of Schizophrenia or schizoaffective disorder
* Clinical diagnosis of Bipolar Affective disorder
* Active suicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
YBOCS Obsessive-Compulsive Severity Score | Bi-monthly (every 2 weeks for duration of trial. Approx. 12 weeks)
  The YBOCS yields an OCD severity score by scoring participants on time, interference, distress, resistance and control of their obsessive and compulsive symptoms on a scale of 0-4. When these scores are summed, they give a total severity score from 0-40. The primary outcome will measure the degree of change in this measurement from pre- to post-treatment.
Clinical Global Improvement - Improvement Scale | Bi-monthly (every 2 weeks for duration of trial. Approx. 12 weeks)
  This is a clinician/Research assistant rated score of clinical improvement. Both treating physician and research assistant (who interviews the participant every two weeks) will independently provide ratings from 1-7, 1 being very much improved and 7 being very much worse.

SECONDARY OUTCOMES:
Change in cortical Inhibition (CI) as measured with Transcranial Magnetic Stimulation. | Pre- and post-treatment (typically, 0 weeks and 12 weeks)
Genotype marker data for SLC1A1, GRIN2B, 5HT1B, 5HT2A and P450 enzymes CYP2D6 and CYP2C19. | Collected at week 0, analyzed periodically (approx. 1x/year)
  We will initially focus on GLU and GABA gene candidates for which there is good evidence of involvement in cortical inhibition. We will also prioritize other markers previously implicated in response and/or etiology of the illness including 5HT1B, 5HT2A, 5HTT, DRD3, DRD4, MOG, BDNF, MAOA, COMT. We will test 200 SNPs across these 12 genes, and also explore any highly promising genes emerging from the literature as time and resources permit. We will test both single markers and haplotypes. Genotyping of CYP2D6 and CYP2C19 will be typed by the Roche Diagnostics Amplichip (www.amplichip.us).
Tolerability/side effects measure with Udvalg for Liniske Undersogelser Side Effect Rating Scale (UKU). | Bi-monthly (every 2 weeks for duration of trial. Approx. 12 weeks)
Clinical Global Impression - Severity Scale. | Bi-monthly (every 2 weeks for duration of trial. Approx. 12 weeks)
Depression symptoms will be rated with the Beck Depression Inventory (BDI). | Bi-monthly (every 2 weeks for duration of trial. Approx. 12 weeks)
DYBOCS (Dimensional Yale-Brown Obsessive-Compulsive Scale) | start, middle and end of trial (typically, 0, 6 and 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Peggy MA Richter, MD FRCPC, Principal Investigator — Sunnybrok Health Sciences Centre; Centre for Addiction and Mental Health; University of Toronto
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Centre for Addiction and Mental Health, Toronto, Ontario